CLINICAL TRIAL: NCT03986645
Title: Clinical Evaluation of 4D Flow Cardiac MRI Sequences - A Prospective Exploratory Study
Brief Title: Clinical Evaluation of 4D Flow Cardiac MRI Sequences
Acronym: Eval-4DFlow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emanuela Valsangiacomo (Other)
Responsible Party: Sponsor-Investigator, Emanuela Valsangiacomo, Prof., University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CIV-16-11-017784
Record Dates: First submitted 2019-05-08; First posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Indication, Unlabeled
Keywords: 4DFlow

STUDY DESIGN:
Intervention Model Description: Prospective, exploratory, non-randomized, interventional study without control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4DFLOW (Experimental): Acquire MR 4DFLow data.
  Interventions: Device: MR data acquisition

INTERVENTIONS:
Device: MR data acquisition — MR data acquisition using CE and non-CE marked pulse sequences.

SUMMARY:
Assess the accuracy of 4D flow cardiac MRI to measure blood flow and velocity, delineate 3D cardiac anatomy and visualize flow dynamics using two (2) different pulse sequences.

DETAILED DESCRIPTION:
Advances in pediatric (cardiac) surgery, interventional techniques and medical care have improved survival for children born with congenital heart disease. Assessment of blood flow and pressures within the heart plays an integral role in the management of patients with congenital or acquired structural heart disease aiding with diagnoses, surveillance for complications, in relation to surgical or catheter procedures, and for therapeutic decision making. Current gold standard, direct intracardiac measurement of flow and pressures is an invasive procedure, while non-invasive echography-Doppler is limited by poor acoustic windows and operator dependency.

Therefore, cardiac MRI (cMRI) has been recommended as an important alternative in imaging of pediatric heart disease. Current clinical standard for MR flow imaging is 2-dimensional providing flow in a single cross-sectional plane. Current clinical CMR protocols in pediatric congenital heart disease are time consuming, depend on technician's experience and require direct supervision by an experienced cardiovascular imaging specialist. 4D Flow is a new approach for cMRI that might overcome these disadvantages. It allows scanning of the entire chest in approximately 7 minutes (depending on field of view, heart rate and resolution). The images can be off-line reconstructed in any plane, avoiding the need to precisely define crosssectional planes during acquisition for each vessel. Owing to time resolved visualizations of intracardiac flow dynamics occult jets or dynamic jets might be more likely to be detected. Potential disadvantages, rsp. potential advantages to be confirmed include lower temporal resolution of 4D sequences than current 2D sequences, unknown consequences of gradient artefacts induced by new velocity encoding schemes and diagnostic plausibility of disease related image features .

ELIGIBILITY:
Inclusion Criteria Patients:

* Clinical referral for cMRI in the absence of any contraindication to cMRI
* Flow measurements are part of the clinical cMRI protocol
* Signed informed consent of participants and/or legal representatives according to current ethical rules and regulations for children and adults
* For females in reproductive age, exclusion of pregnancy by a pregnancy test conducted before the cMRI

Exclusion Criteria Patients:

* Any contraindication for undergoing a cMRI examination or for receiving gadolinium contrast media (renal failure, allergy) per internal institutional policy of University Children's Hospital Zurich
* Any intrathoracic device causing imaging artifacts
* Medical condition at time of examination that would make additional study-related MR scans an unjustified burden or risk.
* Inability or unwillingness to provide informed consent.

Inclusion Criteria Healthy Controls:

* Absence of any contraindication to cMRI
* Signed informed consent of participants according to current ethical rules and regulations
* For females in reproductive age, exclusion of pregnancy by a pregnancy test conducted before the cMRI.

Exclusion Criteria Healthy Controls:

- Any contraindication for undergoing a cMRI examination per internal institutional policy of University Children's Hospital Zurich

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of data processing | Within 72 hours after completion of exam
  Comparison of flow velocities and blood flow measured by 4D flow cMRI pulse sequences against phantom corrected 2D cMRI data.

SECONDARY OUTCOMES:
Image quality | Within 72 hours after completion of exam
  Qualitative grading of 4D flow cMRI anatomical images for image quality using a numerical scale.
Comparability | Within 72 hours after completion of exam
  Qualitative grading of comparability of anatomical findings in 4D flow cMRI anatomical images with contrast-enhanced MR angiography images, if these have been acquired during the clinical examination of patients, using a numerical scale.
Clinical value | Within 72 hours after completion of exam
  Qualitative grading of clinical and diagnostic value of visualizations of flow dynamics using a numerical scale.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Valsangiacomo, Prof. MD, Principal Investigator — UChilldrenZurich